CLINICAL TRIAL: NCT04793906
Title: Meals to Improve Absorption of Iron Supplements and Iron Status in Iron Deficient Women of Reproductive Age: a Randomized, Controlled Trial
Brief Title: Meals to Improve Absorption of Iron Supplements
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Stephen Hennigar, Assistant Professor, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PBRC 2022-036
Record Dates: First submitted 2021-03-03; First posted 2021-03-11 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Iron-deficiency; Iron Deficiency Anemia; Iron Deficiency Anemia Treatment
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — Iron-Dextran Complex

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Beef (Experimental)
  Interventions: Other: Iron supplement with a lunch meal containing beef
- Plant-based alternative (Experimental)
  Interventions: Other: Iron supplement with a lunch meal containing plant-based alternative

INTERVENTIONS:
Other: Iron supplement with a lunch meal containing beef — Participants will consume a lunch meal containing beef with an iron supplement for 8 weeks.
  Arms: Beef
Other: Iron supplement with a lunch meal containing plant-based alternative — Participants will consume a lunch meal containing plant-based alternative with an iron supplement for 8 weeks.
  Arms: Plant-based alternative

SUMMARY:
One of the targeted objectives of Healthy People 2020 is to reduce iron deficiency among women of reproductive age (WRA). Consuming foods rich in iron and/or oral iron supplementation is typically recommended to improve iron status; however, global rates of iron deficiency remain high. Thus, nutritional strategies to improve/maintain iron status are warranted. Dietary iron is found in two different forms: heme and non-heme iron. Non-heme iron is found in plant-based sources and is commonly used as a supplement and food fortificant. Absorption of non-heme iron is low compared to heme iron, which is found in animal sources, such as beef. Studies have also demonstrated that beef contains an unidentified factor that stimulates the absorption of non-heme iron. The primary objective of the proposed study is to determine the effects of incorporating daily meals containing beef or plant-based alternative with or without an iron supplement on indicators of iron status in iron-deficient WRA.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) falls within the normal weight or overweight range (18.5-29.9 kg/m^2)
* Low iron stores (serum ferritin <25 μg/L)
* Willing to refrain from smoking and >2 alcoholic drinks/week for the duration of the study period
* Willing to refrain from vitamin and mineral supplementation for the duration of the study

Exclusion Criteria:

* Currently smoking or vaping
* Currently taking a medication that interferes with micronutrient metabolism
* Unwilling to refrain from vitamin and mineral supplementation for the duration of the study
* Restrictive diets (i.e., vegan or vegetarian diets)
* Metabolic or cardiovascular abnormalities (e.g., kidney disease, diabetes, cardiovascular disease, etc.)
* History of any disease or abnormality of the gastrointestinal tract including, but not limited to, diverticulosis, diverticulitis and inflammatory bowel disease, peptic ulcer disease, Crohn's disease, ulcerative colitis; or previous gastrointestinal surgery
* Blood donation within 4 months of beginning the study
* Abnormal blood clotting

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Assigned Female at birth; identify as a woman
Enrollment: 59 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Iron status | Change from day 0 and day 56
  Plasma ferritin, soluble transferrin receptor, transferrin saturation, hemoglobin and hematocrit will be measured to determine iron status. Changes in measures of iron status during the intervention will be compared between groups.

SECONDARY OUTCOMES:
Profile of Mood States (POMS) | Change from day 0 and day 56
  The POMS questionnaire will be used to assess the overall mood state of the participants. Changes in the POMS during the intervention will be compared between groups.
Appetite | Change from day 0 and day 56
  Subjective appetite and satiety will be assessed before and after the lunch meal using visual analog scales.
Weight | Change from day 0 and day 56
  Changes in body weight during the intervention will be compared between groups.
Body composition | Change from day 0 and day 56
  Body composition (fat mass, fat-free mass, and total body water content) will be determined using single frequency bioimpedance spectroscopy (BIS). Changes in body composition during the intervention will be compared between groups.
Blood pressure | Change from day 0 and day 56
  Changes in blood pressure during the intervention will be compared between groups.
Metabolic biomarkers | Change from day 0 and day 56
  Changes in blood lipids, glucose, and insulin during the intervention will be compared between groups.
Plasma zinc | Change from day 0 and day 56
  Changes in the plasma zinc during the intervention will be compared between groups.
Plasma vitamin B-12 | Change from day 0 and day 56
  Changes in the plasma vitamin B-12 during the intervention will be compared between groups.
Plasma choline | Change from day 0 and day 56
  Changes in the plasma choline during the intervention will be compared between groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hennigar SR, Miller KM, Murphy RD, Braymer A, Mayet CL, Greenway FL, Cheung SN, Weschenfelder C, Berryman CE. Effects of consuming an iron supplement with a meal containing animal or plant-based meat on indicators of iron status and anemia in women of reproductive age with iron deficiency: a randomized, controlled study. Am J Clin Nutr. 2025 Sep;122(3):859-865. doi: 10.1016/j.ajcnut.2025.07.002. Epub 2025 Jul 7. PMID 40633767